CLINICAL TRIAL: NCT01717404
Title: Effects of Mexiletine on Colonic Transit in a Patient With a Known SCN5A A997T Mutation
Brief Title: Effects of Mexiletine on Colonic Transit in a Patient With Irritable Bowel Syndrome - Constipation (IBS-C)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yuri A. Saito Loftus, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-006842
Record Dates: First submitted 2012-10-18; First posted 2012-10-30 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: IBS
Keywords: IBS
MeSH Terms: interventions — Mexiletine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mexiletine (Experimental): 6-day treatment period during which the medication will be taken orally with an initial dose of: 200 mg every 8 hours for 3 doses on day 3, increasing to 300 mg every 8 hours on days 4 and 5 (6 doses), and increasing further to 400 mg every 8 hours on days 6-8 if no telemetry changes and no dose limiting side effects
  Interventions: Drug: Mexiletine

INTERVENTIONS:
Drug: Mexiletine — 6-day treatment period during which the medication will be taken orally with an initial dose of: 200 mg every 8 hours for 3 doses on day 3, increasing to 300 mg every 8 hours on days 4 and 5 (6 doses), and increasing further to 400 mg every 8 hours on days 6-8 if no telemetry changes and no dose limiting side effects

SUMMARY:
To understand if Mexiletine will restores normal colonic motility in a patient with irritable bowel syndrome - constipation (IBS-C) and a genetic mutation in SCN5A.

DETAILED DESCRIPTION:
To understand if Mexiletine will restore normal colonic motility in a patient with a missense mutation in SCN5A, which encodes a voltage-sensitive sodium channel NaV1.5 as it is known to rescue certain expression defects of NaV1.5 in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Established IBS diagnosis with a known A997T mutation in NaV1.5T

Exclusion Criteria:

* Normal 48-hour baseline transit study
* Current use of mexiletine
* Inability to stay in Rochester for 9 days for testing
* Known allergy to mexiletine
* Inability to complete daily diary
* Taking a medication known to affect myotonia, had a coexisting neuromuscular disease, or had another serious medical illness including second- or third-degree heart block, atrial flutter, atrial fibrillation, ventricular arrhythmia, history of cardiac arrhythmia requiring medication, congestive heart failure, symptomatic cardiomyopathy, or symptomatic coronary artery disease
* Inability to withdraw medications known to interact with mexiletine. Patient is currently not on any of these medications

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
change in the 48 hour Colon Transit | Baseline to 10 days
  Colon transit will be measured using validated scintigraphy methods conducted in our Clinical Research Unit (CRU).[17, 18] The participant will ingest a Tc-99m labeled sulfur colloid in egg to be used as a stomach marker and ln-111 chloride bound to activated charcoal enclosed in a methacrylate-coated capsule to measure colonic transit.

CONTACTS AND LOCATIONS:
Overall Officials: Yuri A Saito Loftus, MD, MPH, Principal Investigator — Mayo Clinic

REFERENCES:
- [Derived] Beyder A, Mazzone A, Strege PR, Tester DJ, Saito YA, Bernard CE, Enders FT, Ek WE, Schmidt PT, Dlugosz A, Lindberg G, Karling P, Ohlsson B, Gazouli M, Nardone G, Cuomo R, Usai-Satta P, Galeazzi F, Neri M, Portincasa P, Bellini M, Barbara G, Camilleri M, Locke GR, Talley NJ, D'Amato M, Ackerman MJ, Farrugia G. Loss-of-function of the voltage-gated sodium channel NaV1.5 (channelopathies) in patients with irritable bowel syndrome. Gastroenterology. 2014 Jun;146(7):1659-1668. doi: 10.1053/j.gastro.2014.02.054. Epub 2014 Mar 5. PMID 24613995